CLINICAL TRIAL: NCT02941926
Title: COMPLEEMENT-1: An Open-label, Multicenter, Phase IIIb Study to Assess the Safety and Efficacy of Ribociclib (LEE011) in Combination With Letrozole for the Treatment of Men and Pre/Postmenopausal Women With Hormone Receptor-positive (HR+) HER2-negative (HER2-) Advanced Breast Cancer (aBC) With no Prior Hormonal Therapy for Advanced Disease
Brief Title: Study to Assess the Safety and Efficacy of Ribociclib (LEE011) in Combination With Letrozole for the Treatment of Men and Pre/Postmenopausal Women With HR+ HER2- aBC
Acronym: COMPLEEMENT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A2404; 2016-003467-19 (EudraCT Number); NCT03613220 (obsolete NCT alias)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: HR-positive HER2-negative; advanced breast cancer; LEE011; ribociclib; letrozole; goserelin; CDK; CDK4; CDK6; CDK4/6; Phase IIIb; ER-positive; PR-positive; premenopausal; postmenopausal; men with advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Ribociclib + letrozole+goserelin/leuprolide (Experimental): Participants received ribociclib (orally taken, 3 weeks on/1 week off) in combination with letrozole (orally taken once daily). For men and premenopausal women, either goserelin was given as an injectable subcutaneous implant or leuprolide was given as an intramuscular injection.
  Interventions: Drug: Ribociclib; Drug: Letrozole; Drug: Goserelin; Drug: Leuprolide

INTERVENTIONS:
Drug: Ribociclib — Ribociclib was centrally supplied to the investigators and administered orally once a day on days 1-21 of each 28 day cycle at a starting dose of 600 mg daily
  Other Names: LEE011
Drug: Letrozole — Letrozole was procured locally and administered orally once a day on a continuous daily schedule at a dose of 2.5 mg
Drug: Goserelin — Goserelin was procured locally and administered in men and premenopausal women as an injectable subcutaneous implant administered on day 1 starting at Cycle 1 and then every 28 days at a dose of 3.6 mg (cycle = 28 days)
Drug: Leuprolide — Leuprolide was procured locally and administered in men and premenopausal women as an injectable intramuscular depot administered on day 1 starting at Cycle 1 and then every 28 days at a dose of 7.5 mg (cycle= 28 days)

SUMMARY:
The purpose of this study is to collect additional safety and efficacy data for the combination of ribociclib + letrozole in men and pre/postmenopausal women with HR+HER2- advanced breast cancer and no prior hormonal treatment for advanced disease..

DETAILED DESCRIPTION:
This was an open-label, single arm, multi-center Phase IIIb study. The study was composed of 2 phases: Core Phase and Extension Phase. In the Core Phase, safety and efficacy data was collected. The study treatment during the Core Phase was provided until disease progression, death, unacceptable toxicities, physician's decision, subject/guardian's decision, protocol deviation, study termination by sponsor, lost to follow-up, technical problems or up to 18 months after LPFV.

In the event that patients were still deriving benefit at the end of the Core phase and ribociclib was not approved or available and reimbursed, patients were transitioned to the Extension Phase and continued to receive study treatment until progression, intolerance, death or physician/patient decision. Only safety and clinical benefit (as assessed by investigator) data was collected in the Extension Phase. During the Extension Phase, if ribociclib became locally approved and reimbursed, patients were to be transitioned to prescription. Patients who completed the Extension Phase and continued to derive clinical benefit from the treatment based on the investigator's evaluation received ribociclib from prescription (if approved and reimbursed), another post-trial access program, or other drug access/support program(s).

Canadian sub-study: this sub-study was a multicenter Canadian exploratory correlative sample collection sub-study that aimed to better understand mechanisms of response and resistance to ribociclib in combination with letrozole therapy. This sub-study was available for all Canadian subjects enrolled on the main study and did not alter the planned treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy.
* In the case of women, both pre/perimenopausal and postmenopausal patients were allowed to be included in this study; menopausal status was relevant for the requirement of goserelin to be used concomitantly with ribociclib and letrozole.

  1. Postmenopausal status was defined either by: I).Prior bilateral oophorectomy OR ii). Age ≥ 60 OR iii). Age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and FSH and estradiol in the postmenopausal range per local normal range. If patient was taking tamoxifen or toremifene and age < 60, then FSH and plasma estradiol levels would be in post-menopausal range per local normal range (NCCN Guidelines version 2.2017).

     Note: For women with therapy-induced amenorrhea, serial measurements of FSH and/or estradiol were needed to ensure menopausal status.
  2. Premenopausal status was defined as either: I).Patient had last menstrual period within the last 12 months OR ii). If on tamoxifen or toremifene within the past 14 days, plasma estradiol and FSH must be in the premenopausal range per local normal range OR iii). In case of therapy induced amenorrhea, plasma estradiol and/or FSH must be in the premenopausal range per local normal range.
  3. Perimenopausal status was define as neither premenopausal nor postmenopausal
* Patient had a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory.
* Patient had HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test was required by local laboratory testing.
* Patient had an Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patient had adequate bone marrow and organ function as defined by ALL of the following laboratory values (as assessed by local laboratory):

  * Absolute neutrophil count ≥ 1.5 × 10^9/L
  * Platelets ≥ 100 × 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Potassium, sodium, calcium corrected for serum albumin and magnesium within normal limits or corrected to within normal limits with supplements before first dose of the study medication
  * INR ≤1.5
  * Serum creatinine <1.5 mg/dl or creatinine clearance≥50 mL/min
  * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be below 2.5 × ULN. If the patient had liver metastases, ALT and AST should be < 5 × ULN.
  * Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range in patients with well-documented Gilbert's Syndrome
* Patient must have had a 12-lead ECG with ALL of the following parameters at screening:

  * QTcF interval at screening <450 msec (using Fridericia's correction)
  * Resting heart rate ≥ 50 bpm

Key Exclusion Criteria:

* Patient who received any CDK4/6 inhibitor
* Patient who received any prior systemic hormonal therapy for advanced breast cancer; no more than one prior regimen of chemotherapy for the treatment of metastatic disease was permitted. Note:

  * Patients who received (neo) adjuvant therapy for breast cancer were eligible. If the prior neo (adjuvant) therapy included letrozole or anastrozole the disease free interval had to be greater than 12 months from the completion of treatment until study entry.
  * Patients who received ≤ 28 days of letrozole or anastrozole for advanced disease prior to inclusion in this trial were eligible.
  * Any prior (neo) adjuvant anti-cancer therapy or prior chemotherapy for metastatic disease had to be stopped at least 5 half-lives or 7 days, whichever was longer, before study inclusion.
* Patient was concurrently using other anti-cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3246 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (429):
- United States (71):
  - Alaska Cancer Research and Education Center, Anchorage, Alaska
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Arizona Oncology Associates, Phoenix, Arizona
  - Arizona Oncology Associates Arizona Oncology Assoc. (2), Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Pacific Shores Medical Group SC, Long Beach, California
  - USC Norris Cancer Center, Los Angeles, California
  - University of California Irvine UC Irvine (11), Orange, California
  - Ventura County Hematology and Oncology, Oxnard, California
  - PCR Oncology, Pismo Beach, California
  - California Pacific Medical Center Onc Dept, San Francisco, California
  - Centura Health Research Center Centura Health Research Center, Denver, Colorado
  - Poudre Valley Hospital Poudre Valley Health System, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Florida Cancer Research Institute Dept of Oncology, Davie, Florida
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Watson Clinic Center for Research 1730 Location, Lakeland, Florida
  - Mid Florida Hematology and Onc Ctr, Orange, Florida
  - Summit Cancer Care Summit Cancer Care (SC), Savannah, Georgia
  - John D Archbold Memorial Hospital John D. Archbold Mem Hosp (4), Thomasville, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Stroger Cook County Hospital Division of Hematology & Onc, Chicago, Illinois
  - Joliet Oncology-Hematology Associates Presence Cancer Center, Joliet, Illinois
  - Mid Illinois Hematology Oncology Mid Illinois Hema/Onc (3), Normal, Illinois
  - Alpha Med Physician Group, LLC, Tinley Park, Illinois
  - Indian Univ Health Goshen Center forCancer SC, Goshen, Indiana
  - Northwest Oncology, Munster, Indiana
  - June E. Nylan Cancer Center, Sioux City, Iowa
  - University of Kansas Medical Center University of Kansas Med Ctr 9, Kansas City, Kansas
  - Sarah Cannon at Overland Park Regional Medical Center, Overland Park, Kansas
  - John Ochsner Heart and Vascular Institute Clinical Trials, New Orleans, Louisiana
  - Northern Light Mercy Hospital SC, Portland, Maine
  - Greater Baltimore Medical Center Cancer Center Greater Baltimore Medical Ctr, Baltimore, Maryland
  - Maryland Oncology Hematology P A Columbia, Rockville, Maryland
  - Kaiser Permanente, Rockville, Maryland
  - Medical Faculty Assc Inc Medical Faculty Assc., Inc. (2, Washington DC, Maryland
  - Jackson Oncology Associates, Jackson, Mississippi
  - Nebraska Hematology-Oncology, P.C., Lincoln, Nebraska
  - Nebraska Cancer Specialists Oncology Hematology West, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada CCC of Nevada Henderson (4), Henderson, Nevada
  - Trinitas Comprehensive Cancer Center, Elizabeth, New Jersey
  - Englewood Health, Englewood, New Jersey
  - The Valley Hospital / Luckow Pavillion, Paramus, New Jersey
  - Somerset Hematology Oncology Associates Somerset Hematolgy Onc -MI, Somerset, New Jersey
  - New Mexico Cancer Care Alliance ., Albuquerque, New Mexico
  - San Juan Oncology Associates, Farmington, New Mexico
  - Clinical Research Alliance, Lake Success, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Oncology Speciialists of Charlotte, Charlotte, North Carolina
  - Aultman Cancer Center Main Centre, Canton, Ohio
  - The Christ Hospital Cancer Center Research Program Linder Research Center, Cincinnati, Ohio
  - University Hospitals of Cleveland Seidman Cancer Center Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation Cleveland Clinic (5), Cleveland, Ohio
  - Dayton Physicians, Kettering, Ohio
  - Oklahoma Cancer Specialists and Research Institute SC-2, Tulsa, Oklahoma
  - Oregon Health Sciences University SC-5, Portland, Oregon
  - McLeod Center for Cancer Treatment and Research, Florence, South Carolina
  - Carolina Blood and Cancer Care of South Carolina, Rock Hill, South Carolina
  - Millennium Research Clin Develop Millennium Oncology - FL, Houston, Texas
  - Mays Cancer Ctr Uthsa Mdacc, San Antonio, Texas
  - Hope Cancer Center of East Texas, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - PeaceHealth St Joseph Medical Center, Bellingham, Washington
  - Providence Regional Medical Centre of Everett, Everett, Washington
  - Kadlec Clinic Hematology and Onco, Kennewick, Washington
  - Valley Medical Center Research Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center-Oncology SC, Seattle, Washington
  - Northwest Medical Specialties Dept.ofNW Med. Specialties, Tacoma, Washington
  - Columbia St Mary s Hospital of Milwaukee St. Mary's Hospital Ozaukee, Milwaukee, Wisconsin
  - Cheyenne Regional Medical Center Cheyenne Regional Med Ctr (3), Cheyenne, Wyoming
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, La Rioja
- Austria (6):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (18):
  - Novartis Investigative Site, Luxembourg, Luxembourg
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Mons
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Wilrijk
- Bulgaria (3):
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (28):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Sault Ste. Marie, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, Santiago, Chile
- Czechia (10):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Vejle
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Oulu
  - Novartis Investigative Site, Tampere
- France (37):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Tours, Indre Et Loire
  - Novartis Investigative Site, Reims, Marne
  - Novartis Investigative Site, Albi
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Mont-de-Marsan
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Périgueux
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Plerin Sur Mer
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulon La Seyne Sur Mer
  - Novartis Investigative Site, Troyes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Greece (5):
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Hong Kong (3):
  - Novartis Investigative Site, Pokfulam, Hong Kong
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- India (11):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Tamil Nadu, Chennai
  - Novartis Investigative Site, Admedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi
- Israel (6):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (60):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Asti, AT
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Benevento, BN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Monserrato, CA
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Grosseto, GR
  - Novartis Investigative Site, Lecco, LC
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Lucca, LU
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Taormina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Nuoro, NU
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Fano, PU
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Savona, SV
  - Novartis Investigative Site, Trento, TN
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Saronno, VA
  - Novartis Investigative Site, Mirano, VE
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Viterbo, VT
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
- Novartis Investigative Site, Amman, Jordan
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Malaysia (5):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Putrajaya, Kuala Lumpur
  - Novartis Investigative Site, Tanjong Bungah, Pulau Pinang
  - Novartis Investigative Site, Petaling Jaya, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (2):
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mexico City
- Netherlands (24):
  - Novartis Investigative Site, Maastricht, AZ
  - Novartis Investigative Site, Venray, CE
  - Novartis Investigative Site, Apeldoorn, DZ
  - Novartis Investigative Site, Arnhem, Gelderland
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Beverwijk
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Goes
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Hilversum
  - Novartis Investigative Site, Hoofddorp
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Roermond
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Zutphen
  - Novartis Investigative Site, Zwolle
- Norway (3):
  - Novartis Investigative Site, Grålum
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Stavanger
- Novartis Investigative Site, Muscat, Oman
- Novartis Investigative Site, Panama City, Panama
- Philippines (3):
  - Novartis Investigative Site, City of Taguig, National Capital Region
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, San Juan City
- Poland (10):
  - Novartis Investigative Site, Żory, Silesian Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (4):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (14):
  - Novartis Investigative Site, Leningrad Region, Russia
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Kaluga
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Moscow Region Istra Village
  - Novartis Investigative Site, Moscow Rerion Balashiha
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yaroslavl
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Mecca
  - Novartis Investigative Site, Riyadh
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Poprad
- Slovenia (2):
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Maribor
- Spain (40):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canarias, Las Palmas de Gran Canaria
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Reus, Tarragona
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Castellon, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Granollers
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Sweden (5):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Vaxjo
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Thailand (4):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (26):
  - Novartis Investigative Site, Peterborough, Cambridgeshire
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Portsmouth, Hants
  - Novartis Investigative Site, Maidstone, Kent
  - Novartis Investigative Site, York, North Yorkshire
  - Novartis Investigative Site, Aberdeen, Scotland
  - Novartis Investigative Site, Ipswich, Suffolk
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, East Sussex
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] Caputo R, Fabi A, Romagnoli E, Baldini E, Grasso D, Fenderico N, Michelotti A. Ribociclib Plus Letrozole in Italian Male Patients with Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Case Studies of Phase 3b CompLEEment-1 Trial. Breast Cancer (Dove Med Press). 2022 Oct 18;14:351-362. doi: 10.2147/BCTT.S376902. eCollection 2022. PMID 36267663
- [Derived] Salvador Bofill J, Moreno Anton F, Rodriguez Sanchez CA, Galve Calvo E, Hernando Melia C, Ciruelos Gil EM, Vidal M, Jimenez-Rodriguez B, De la Cruz Merino L, Martinez Janez N, Villanueva Vazquez R, de Toro Salas R, Anton Torres A, Alvarez Lopez IM, Gavila Gregori J, Quiroga Garcia V, Vicente Rubio E, De la Haba-Rodriguez J, Gonzalez-Santiago S, Diaz Fernandez N, Barnadas Molins A, Cantos Sanchez de Ibarguen B, Delgado Mingorance JI, Bellet Ezquerra M, de Casa S, Gimeno A, Martin M. Safety and efficacy of ribociclib plus letrozole in patients with HR+, HER2- advanced breast cancer: Results from the Spanish sub-population of the phase 3b CompLEEment-1 trial. Breast. 2022 Dec;66:77-84. doi: 10.1016/j.breast.2022.09.006. Epub 2022 Sep 28. PMID 36206609
- [Derived] De Laurentiis M, Caputo R, Mazza M, Mansutti M, Masetti R, Ballatore Z, Torrisi R, Michelotti A, Zambelli A, Ferro A, Generali D, Vici P, Coltelli L, Fabi A, Marchetti P, Ballestrero A, Spazzapan S, Frassoldati A, Sarobba MG, Grasso D, Zamagni C. Safety and Efficacy of Ribociclib in Combination with Letrozole in Patients with HR+, HER2- Advanced Breast Cancer: Results from the Italian Subpopulation of Phase 3b CompLEEment-1 Study. Target Oncol. 2022 Nov;17(6):615-625. doi: 10.1007/s11523-022-00913-x. Epub 2022 Sep 24. PMID 36152144
- [Derived] Campone M, De Laurentiis M, Zamagni C, Kudryavcev I, Agterof M, Brown-Glaberman U, Palacova M, Chatterjee S, Menon-Singh L, Wu J, Martin M. Ribociclib plus letrozole in male patients with hormone receptor-positive, human epidermal growth factor receptor 2-negative advanced breast cancer: subgroup analysis of the phase IIIb CompLEEment-1 trial. Breast Cancer Res Treat. 2022 May;193(1):95-103. doi: 10.1007/s10549-022-06543-1. Epub 2022 Feb 25. PMID 35212906
- [Derived] De Laurentiis M, Borstnar S, Campone M, Warner E, Bofill JS, Jacot W, Dent S, Martin M, Ring A, Cottu P, Lu J, Ciruelos E, Azim HA, Chatterjee S, Zhou K, Wu J, Menon-Singh L, Zamagni C. Full population results from the core phase of CompLEEment-1, a phase 3b study of ribociclib plus letrozole as first-line therapy for advanced breast cancer in an expanded population. Breast Cancer Res Treat. 2021 Oct;189(3):689-699. doi: 10.1007/s10549-021-06334-0. Epub 2021 Aug 19. PMID 34414532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Core Phase was conducted across 514 centers in 38 countries. Extension Phase was conducted across 189 centers in 25 countries.
Pre-assignment Details: A total of 3694 participants were screened in this study of which 3246 participants were enrolled in the study.
Groups:
- Ribociclib + Letrozole + Goserelin/Leuprolide: Participants received ribociclib (orally taken, 3 weeks on/1 week off) in combination with letrozole (orally taken once daily). For men and premenopausal women, either goserelin was given as an injectable subcutaneous implant or leuprolide was given as an intramuscular injection.
Period: Core Phase
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Started | 3246
Canadian Sub-study (Participants who participated in the Canadian sub-study) | 88
Completed | 1301
Not Completed | 1945
Not completed — Progressive disease | 1109
Not completed — Adverse Event | 504
Not completed — Subject/guardian decision | 127
Not completed — Physician Decision | 112
Not completed — Death | 46
Not completed — Protocol deviation | 34
Not completed — Lost to Follow-up | 8
Not completed — Technical problems | 5
Period: Extension Phase
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Started (Subjects from countries where ribociclib was not yet approved and reimbursed who were still deriving benefit at the end of the Core Phase) | 413
Completed | 112
Not Completed | 301
Not completed — Physician Decision | 155
Not completed — Progressive disease | 115
Not completed — Adverse Event | 13
Not completed — Subject/Guardian decision | 12
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 3246
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3207
  Male | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2553
  Unknown | 284
  Asian | 227
  Other | 134
  Black | 29
  Native American | 18
  Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) During Treatment With Ribociclib + Letrozole in the Core Phase
Description: AEs were defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s).
  SAEs were defined as meeting at least 1 of the following criteria: is fatal or life-threatening, Results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, is medically significant, requires inpatient hospitalization or prolongation of existing hospitalization. A SAE which caused death of the participant was considered as fatal SAE.
  AEs were assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1 to 5 were used to characterize the severity of the Adverse Event. Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening and Grade 5: death related to AE.
  A participant with multiple severity grades for an AE is only counted under the maximum grade.
Time Frame: From start of treatment up to 30 days after last treatment (for participants who did not enter to the Extension phase) or up to last treatment in the Core phase (for participants who entered the Extension phase), assessed up to approximately 33 months.
Population: Safety set in the Core phase: All participants who received at least one dose of study treatment defined as either ribociclib, or letrozole, or goserelin, or leuprolide in the Core phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 3246
Participants
  AEs- All grades | 3203
  AEs- Grade ≥ 3 | 2461
  Treatment-related AEs- All grades | 3091
  Treatment-related AEs- Grade ≥ 3 | 2192
  SAEs- All grades | 702
  SAEs- Grade ≥ 3 | 590
  Treatment-related SAEs- All grades | 203
  Treatment-related SAEs- Grade ≥ 3 | 178
  Fatal SAEs- All grades | 62
  Treatment-related Fatal SAEs- All grades | 14
  AEs leading to discontinuation- All grades | 528
  AEs leading to discontinuation- Grade ≥ 3 | 310
  Treatment-related AEs leading to discontinuation- All grades | 418
  Treatment-related AEs leading to discontinuation-Grade ≥ 3 | 237
  AEs leading to dose adjustment/interruption- All grades | 2434
  AEs leading to dose adjustment/interruption- Grade ≥ 3 | 2095
  Treatment-related AEs leading to dose adjustment/interruption- All grades | 2235
  Treatment-related AEs leading to dose adjustment/interruption- Grade ≥ 3 | 1964
  AEs requiring additional therapy- All grades | 2624
  AEs requiring additional therapy- Grade ≥ 3 | 844
  Treatment-related AEs requiring additional therapy- All grades | 1613
  Treatment-related AEs requiring additional therapy- Grade ≥ 3 | 392

2. Secondary Outcome: Time-to-Progression (TTP) Based on Investigator's Assessment (Core Phase)
Description: Time to progression (TTP) is defined as time from date of start of treatment to the date of first documented progression or death due to underlying cancer. Participants with symptoms of rapidly progressing disease without radiologic evidence were classified as progression only when clear evidence of clinical deterioration was documented and/or patient discontinued due to 'Disease progression' or death due to study indication. When there was no documentation of radiologic evidence of progression, and the patient discontinued for 'Disease progression' due to documented clinical deterioration of disease, the date of discontinuation was used as date of progression.
  TTP was estimated using the Kaplan-Meier method. 95% CI of median was calculated according to Brookmeyer and Crowley method.
Time Frame: Up to approximately 33 months
Population: Full Analysis set: All participants who received at least one dose of study treatment defined as either ribociclib, or letrozole, or goserelin, or leuprolide in the Core phase.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 3246
Months | 27.1 [25.7 to NA] — Upper limit was not reached (NA) due to insufficient follow up time

3. Secondary Outcome: Overall Response Rate (ORR) Based on Investigator's Assessment (Core Phase)
Description: Overall response rate (ORR) is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 based on investigator's assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  95% CI was calculated using the exact binomial method.
Time Frame: Up to approximately 33 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 3246
Percentage of participants | 29.3 [27.7 to 30.9]

4. Secondary Outcome: Clinical Benefit Rate (CBR) Based on Investigator's Assessment (Core Phase)
Description: Clinical benefit rate (CBR) is defined as the percentage of participants with a best overall response of complete response (CR), or partial response (PR) or an overall lesion response of stable disease (SD), lasting as per local review, for a duration of at least 24 weeks. CR, PR and SD are defined according to RECIST 1.1 based on investigator's assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
  95% CI was calculated using the exact binomial method.
Time Frame: Up to approximately 33 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 3246
Percentage of participants | 70.7 [69.1 to 72.2]

5. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Breast (FACT-B) Score (Core Phase)
Description: Change from baseline in FACT-B scores was assessed. FACT-B is a self-report instrument that measures multidimensional quality of life (QOL) in patients with breast cancer. The FACT-B consists of 37 questions that address physical, social, emotional, and functional well-being, with specific questions relevant to women with breast cancer. Each item has a score range of 0 (Not at all) to 4 (Very much), with a total score ranging from 0-148. The higher the score, the better the QOL reported by the participant. A positive change from baseline indicates improvement in QoL.
  Due to the nature of the questionnaire, only females were asked to complete this questionnaire.
Time Frame: On Day 1 of Cycle 1, 2, 3, 4 ,5, 6, 8, 10, 12 and after that every 3 cycles, and End of treatment, assessed up to 33 months. Cycle=28 days
Population: Female participants in the Full Analysis set population for whom baseline and at least one post baseline patient-reported outcome measurements are available. Number analyzed indicates number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 1230
Score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 1100
  Cycle 2 Day 1 | 0.2 (13.29)
  Cycle 3 Day 1: number analyzed (Participants) | 993
  Cycle 3 Day 1 | 0.1 (13.72)
  Cycle 4 Day 1: number analyzed (Participants) | 884
  Cycle 4 Day 1 | -0.3 (14.90)
  Cycle 5 Day 1: number analyzed (Participants) | 852
  Cycle 5 Day 1 | 0.0 (15.02)
  Cycle 6 Day 1: number analyzed (Participants) | 839
  Cycle 6 Day 1 | -0.8 (14.91)
  Cycle 8 Day 1: number analyzed (Participants) | 726
  Cycle 8 Day 1 | -0.9 (16.32)
  Cycle 10 Day 1: number analyzed (Participants) | 683
  Cycle 10 Day 1 | -1.2 (15.83)
  Cycle 12 Day 1: number analyzed (Participants) | 680
  Cycle 12 Day 1 | -1.6 (16.13)
  Cycle 15 Day 1: number analyzed (Participants) | 602
  Cycle 15 Day 1 | -2.0 (16.58)
  Cycle 18 Day 1: number analyzed (Participants) | 538
  Cycle 18 Day 1 | -2.0 (16.09)
  Cycle 21 Day 1: number analyzed (Participants) | 473
  Cycle 21 Day 1 | -2.0 (17.82)
  Cycle 24 Day 1: number analyzed (Participants) | 289
  Cycle 24 Day 1 | -3.0 (17.89)
  Cycle 27 Day 1: number analyzed (Participants) | 145
  Cycle 27 Day 1 | -2.7 (13.84)
  Cycle 30 Day 1: number analyzed (Participants) | 32
  Cycle 30 Day 1 | -2.0 (14.14)
  Cycle 33 Day 1: number analyzed (Participants) | 2
  Cycle 33 Day 1 | 12.1 (21.10)
  End of Treatment: number analyzed (Participants) | 861
  End of Treatment | -4.1 (16.98)

6. Secondary Outcome: Number of Participants With AEs and SAEs in the Extension Phase
Description: AEs were defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s).
  SAEs were defined as meeting at least 1 of the following criteria: is fatal or life-threatening, Results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, is medically significant, requires inpatient hospitalization or prolongation of existing hospitalization.
  AEs were assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1 to 5 were used to characterize the severity of the Adverse Event. Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening and Grade 5: death related to AE.
  A participant with multiple severity grades for an AE is only counted under the maximum grade.
Time Frame: From first dose of treatment in the Extension phase up to 30 days after last dose of treatment, assessed up approximately 37.6 months
Population: Safety set in the Extension phase: all patients who received at least one dose of study medications defined as ribociclib or letrozole or goserelin/leuprolide (if applicable) in the Extension Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 413
Participants
  AEs- All grades | 297
  AEs- Grade ≥ 3 | 159
  Treatment-related AEs- All grades | 221
  Treatment-related AEs- Grade ≥ 3 | 123
  SAEs- All grades | 54
  SAEs- Grade ≥ 3 | 45
  Treatment-related SAEs- All grades | 7
  Treatment-related SAEs- Grade ≥ 3 | 6
  Fatal SAEs- All grades | 5
  Treatment-related Fatal SAEs- All grades | 0
  AEs leading to discontinuation- All grades | 17
  AEs leading to discontinuation- Grade ≥ 3 | 9
  Treatment-related AEs leading to discontinuation- All grades | 7
  Treatment-related AEs leading to discontinuation-Grade ≥ 3 | 4
  AEs leading to dose adjustment/interruption- All grades | 185
  AEs leading to dose adjustment/interruption- Grade ≥ 3 | 132
  Treatment-related AEs leading to dose adjustment/interruption- All grades | 134
  Treatment-related AEs leading to dose adjustment/interruption- Grade ≥ 3 | 113
  AEs requiring additional therapy- All grades | 186
  AEs requiring additional therapy- Grade ≥ 3 | 56
  Treatment-related AEs requiring additional therapy- All grades | 47
  Treatment-related AEs requiring additional therapy- Grade ≥ 3 | 12

7. Secondary Outcome: Number of Participants With Clinical Benefit (Extension Phase)
Description: Clinical benefit as assessed by the Investigator during Extension phase
Time Frame: On Day 1 of every 3 cycles, starting from Cycle 1 of the Extension phase until end of treatment, assessed up to 37.4 months. Cycle= 28 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 413
Participants
  Cycle 1 Day 1 | 413
  Cycle 4 Day 1 | 386
  Cycle 7 Day 1 | 353
  Cycle 10 Day 1 | 323
  Cycle 13 Day 1 | 245
  Cycle 16 Day 1 | 200
  Cycle 19 Day 1 | 183
  Cycle 22 Day 1 | 118
  Cycle 25 Day 1 | 55
  Cycle 28 Day 1 | 51
  Cycle 31 Day 1 | 44
  Cycle 34 Day 1 | 32
  Cycle 37 Day 1 | 24
  Cycle 40 Day 1 | 5

8. Other Pre Specified Outcome: Canadian Sub-study: Proteomic Analysis of Ribociclib and Letrozole Cohort Not Achieving Clinical Benefit Compared to a Cohort Sensitive to Treatment With Ribociclib and Letrozole
Description: Exploratory analysis performed in archival tumor samples collected during screening in the main study. Protein expression levels of the ribociclib plus letrozole cohort that did not achieve clinical benefit (progression within 3 months of treatment) and the cohort sensitive to ribociclib and letrozole (cohort with a time to progression of 22 months or more) were determined using using Single-Pot, Solid-Phase-enhanced, Sample Preparation-Clinical Tissue Proteomics (SP3-CTP). For normalization purposes a pooled internal standard sample, comprised of aliquots of every sample included in the study, was included in each experimental batch. Protein abundances were calculated as the log2 transformed abundances relative to the pooled internal standard. Positive values represent higher protein expression levels compared to the pooled internal standard. Expression levels of proteins that showed association to predicting response to study treatment are presented.
Time Frame: Screening (up to 28 days before first dose of study treatment)
Population: Participants included in the sub-study (only available for Canadian participants) with evaluable tumor samples collected during screening in the main study and with time to progression within 3 months (cohort not achieving clinical benefit) or with time to progression of 22 months or more (cohort sensitive to treatment)
Measure: Mean (Standard Deviation); unit: log2 transformed relative ratio
Groups:
- Primary Resistance Cohort: Participants included in the sub-study treated with ribociclib in combination with letrozole and goserelin or leuprolide (for men and premenopausal women) who did not achieve clinical benefit (tumor progressed within 3 months of treatment)
- Sensitive Cohort: Participants included in the sub-study treated with ribociclib in combination with letrozole and goserelin or leuprolide (for men and premenopausal women) who were sensitive to treatment (with time to progression of 22 months or more)
Arm/Group | Primary Resistance Cohort | Sensitive Cohort
Number analyzed (Participants) | 8 | 19
log2 transformed relative ratio
  Isocitrate dehydrogenase [NADP] cytoplasmic (IDH1) | 0.112 (0.500) | -0.218 (0.352)
  Retinal dehydrogenase 1 (ALDH1A1) | 0.022 (0.446) | -0.325 (0.147)
  Coagulation factor XIII A chain (F13A1) | -0.378 (0.263) | -0.010 (0.198)
  Argininosuccinate synthase (ASS1) | 0.104 (0.612) | -0.466 (0.129)
  Heat shock protein beta-1 (HSPB1) | -0.546 (0.113) | -0.151 (0.270)
  Aldehyde dehydrogenase, mitochondrial (ALDH2) | 0.319 (0.571) | -0.077 (0.374)
  Decorin (DCN) | -0.456 (0.266) | -0.033 (0.568)
  Cathepsin G (CTSG) | -0.634 (0.191) | -0.175 (0.274)
  Pyruvate carboxylase, mitochondrial (PC) | 0.413 (0.649) | -0.004 (0.181)
  C-1-tetrahydrofolate synthase, cytoplasmic (MTHFD1) | 0.033 (0.254) | -0.129 (0.087)
  Collagen alpha-3(VI) chain (COL6A3) | -0.186 (0.187) | -0.015 (0.186)
  Versican core protein (VCAN) | -0.301 (0.242) | 0.141 (0.581)
  Fibulin-1 (FBLN1) | -0.245 (0.313) | 0.128 (0.435)
  Acetyl-CoA acetyltransferase, mitochondrial (ACAT1) | 0.135 (0.409) | -0.074 (0.136)
  Long-chain-fatty-acid--CoA ligase 1 (ACSL1) | 0.296 (1.056) | -0.144 (0.205)
  Pigment epithelium-derived factor (SERPINF1) | -0.378 (0.161) | 0.169 (0.662)
  3-ketoacyl-CoA thiolase, mitochondrial (ACAA2) | 0.258 (0.501) | -0.080 (0.166)
  Fatty acid synthase (FASN) | -0.198 (0.198) | 0.038 (0.284)
  Lumican (LUM) | -0.355 (0.182) | 0.010 (0.399)
  Fibulin-2 (FBLN2) | -0.208 (0.098) | 0.075 (0.271)
  Prolow-density lipoprotein receptor-related protein 1 (LRP1) | -0.148 (0.118) | 0.094 (0.194)
  Galectin-3-binding protein (LGALS3BP) | -0.491 (0.134) | -0.126 (0.213)
  Inactive tyrosine-protein kinase 7 (PTK7) | -0.251 (0.071) | 0.070 (0.237)
  Ras GTPase-activating-like protein IQGAP2 (IQGAP2) | 0.318 (0.538) | -0.036 (0.221)
  Spectrin alpha chain, non-erythrocytic 1 (SPTAN1) | 0.085 (0.323) | -0.082 (0.123)
  Periostin (POSTN) | -0.419 (0.165) | 0.051 (0.393)
  Procollagen C-endopeptidase enhancer 1 (PCOLCE) | -0.217 (0.172) | 0.184 (0.375)
  CD109 antigen (CD109) | -0.213 (0.141) | 0.043 (0.145)
  Palladin (PALLD) | -0.207 (0.137) | 0.050 (0.221)
  Collagen triple helix repeat-containing protein 1 (CTHRC1) | -0.514 (0.156) | 0.176 (0.387)
  Collagen alpha-1(XII) chain (COL12A1) | -0.302 (0.183) | 0.230 (1.041)
  Matrix-remodeling-associated protein 5 (MXRA5) | -0.221 (0.192) | 0.205 (0.431)
  C-type mannose receptor 2 (MRC2) | -0.201 (0.124) | 0.170 (0.274)

9. Post Hoc Outcome: All Collected Deaths
Description: On-treatment- Core phase: from first treatment in the Core phase up to 30 days post-treatment (for participants who did not enter the Extension phase) or up to last treatment in the Core phase (for participants who entered the Extension phase). Extension phase: from first dose of treatment in the Extension phase up to 30 days after last dose of treatment.
  Post-treatment survival follow-up- Core phase: from 31 days post-treatment in the core phase up to end of study; Extension phase: from 31 days post-treatment in the Extension phase up to end of study.
Time Frame: On-treatment Core Phase: up to 33 months; Post-treatment survival Follow-up Core Phase: Up to 33 months; On-treatment Extension Phase: up to approximately 37.6 months; Post-treatment survival Follow-up Extension Phase: Up to approximately 37.6 months.
Population: Core phase: All participants who received at least one dose of study treatment defined as either ribociclib, or letrozole, or goserelin, or leuprolide in the Core phase.
  Extension phase: all patients who received at least one dose of study medications defined as ribociclib or letrozole or goserelin/leuprolide (if applicable) in the Extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib + Letrozole + Goserelin/Leuprolide
Number analyzed (Participants) | 3246
Participants
  On-treatment Core Phase | 74
  Post-treatment survival follow-up Core Phase: number analyzed (Participants) | 2759
  Post-treatment survival follow-up Core Phase | 90
  All deaths Core Phase | 164
  On-treatment Extension Phase: number analyzed (Participants) | 413
  On-treatment Extension Phase | 5
  Post-treatment survival follow-up Extension Phase: number analyzed (Participants) | 408
  Post-treatment survival follow-up Extension Phase | 3
  All deaths Extension Phase: number analyzed (Participants) | 413
  All deaths Extension Phase | 8

ADVERSE EVENTS:
Time Frame: On-treatment-Core phase: from first treatment to 30 days post-treatment or last treatment in the Core phase (for extension phase participants), up to 33 months; Extension phase: from first treatment in the Extension phase to 30 days post-treatment, up to approx. 37.6 months.Post-treatment survival-Core phase: from 31 days post-treatment in the Core phase to study end, up to 33 months; Extension phase: from 31 days post-treatment in the Extension phase up to study end, up to approx.. 37.6 months.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment follow-up period are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period
Groups:
- All Patients- On-treatment Core Phase: AEs collected in the on-treatment period of the core phase (up to 30 days after last treatment for participants who did not enter the Extension phase or up to last treatment in the Core phase for participants who entered the Extension phase)
- All Patients- On-treatment Extension Phase: AEs collected in the on-treatment period of the Extension phase (from first dose of treatment in the Extension phase up to 30 days after last dose of treatment)
- All-patients- Post-treatment Survival Follow-up Core Phase: Deaths collected in the post-treatment survival follow-up period (starting from 31 days post-treatment in the Core phase). No AEs were collected during this period
- All-patients- Post-treatment Survival Follow-up Extension Phase: Deaths collected in the post-treatment survival follow-up period (starting from 31 days post-treatment in the Extension phase). No AEs were collected during this period
Arm/Group | All Patients- On-treatment Core Phase | All Patients- On-treatment Extension Phase | All-patients- Post-treatment Survival Follow-up Core Phase | All-patients- Post-treatment Survival Follow-up Extension Phase
All-Cause Mortality (participants affected / at risk) | 74/3246 | 5/413 | 90/2759 | 3/408
Serious Adverse Events (participants affected / at risk) | 702/3246 | 54/413 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3150/3246 | 247/413 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients- On-treatment Core Phase (N=3246) | All Patients- On-treatment Extension Phase (N=413) | All-patients- Post-treatment Survival Follow-up Core Phase (N=0) | All-patients- Post-treatment Survival Follow-up Extension Phase (N=0)
Anaemia (Blood and lymphatic system disorders) | 24 | 0 | NA | NA
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 0 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | NA | NA
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 9 | 0 | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0 | NA | NA
Acute coronary syndrome (Cardiac disorders) | 3 | 0 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | NA | NA
Angina pectoris (Cardiac disorders) | 2 | 0 | NA | NA
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | NA | NA
Arrhythmia (Cardiac disorders) | 1 | 0 | NA | NA
Atrial fibrillation (Cardiac disorders) | 7 | 0 | NA | NA
Atrial flutter (Cardiac disorders) | 1 | 0 | NA | NA
Atrioventricular block (Cardiac disorders) | 1 | 0 | NA | NA
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | NA | NA
Bradycardia (Cardiac disorders) | 1 | 0 | NA | NA
Cardiac arrest (Cardiac disorders) | 3 | 1 | NA | NA
Cardiac disorder (Cardiac disorders) | 1 | 0 | NA | NA
Cardiac failure (Cardiac disorders) | 3 | 0 | NA | NA
Cardiac failure acute (Cardiac disorders) | 1 | 0 | NA | NA
Cardiac failure congestive (Cardiac disorders) | 3 | 0 | NA | NA
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | NA | NA
Cor pulmonale (Cardiac disorders) | 1 | 0 | NA | NA
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | NA | NA
Myocardial infarction (Cardiac disorders) | 5 | 0 | NA | NA
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | NA | NA
Palpitations (Cardiac disorders) | 1 | 0 | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | NA | NA
Ventricular dysfunction (Cardiac disorders) | 1 | 0 | NA | NA
Vertigo (Ear and labyrinth disorders) | 2 | 0 | NA | NA
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | NA | NA
Amaurosis fugax (Eye disorders) | 1 | 0 | NA | NA
Cataract (Eye disorders) | 1 | 0 | NA | NA
Eyelid ptosis (Eye disorders) | 1 | 0 | NA | NA
Keratitis (Eye disorders) | 1 | 0 | NA | NA
Retinal detachment (Eye disorders) | 1 | 0 | NA | NA
Ulcerative keratitis (Eye disorders) | 1 | 0 | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 16 | 1 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | NA | NA
Ascites (Gastrointestinal disorders) | 4 | 0 | NA | NA
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Colitis (Gastrointestinal disorders) | 3 | 0 | NA | NA
Constipation (Gastrointestinal disorders) | 6 | 0 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 14 | 0 | NA | NA
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | NA | NA
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 1 | NA | NA
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0 | NA | NA
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastritis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | NA | NA
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | NA | NA
Ileus (Gastrointestinal disorders) | 2 | 0 | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 6 | 0 | NA | NA
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | NA | NA
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 12 | 0 | NA | NA
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | NA | NA
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | NA | NA
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | NA | NA
Rectal stenosis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | NA | NA
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0 | NA | NA
Stomatitis (Gastrointestinal disorders) | 2 | 0 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 31 | 2 | NA | NA
Adverse drug reaction (General disorders) | 1 | 0 | NA | NA
Asthenia (General disorders) | 6 | 0 | NA | NA
Chest discomfort (General disorders) | 1 | 0 | NA | NA
Chills (General disorders) | 1 | 0 | NA | NA
Death (General disorders) | 1 | 0 | NA | NA
Disease progression (General disorders) | 1 | 0 | NA | NA
Fatigue (General disorders) | 5 | 0 | NA | NA
Gait disturbance (General disorders) | 2 | 0 | NA | NA
General physical health deterioration (General disorders) | 13 | 0 | NA | NA
Influenza like illness (General disorders) | 1 | 0 | NA | NA
Infusion site extravasation (General disorders) | 1 | 0 | NA | NA
Localised oedema (General disorders) | 1 | 0 | NA | NA
Malaise (General disorders) | 3 | 0 | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | NA | NA
Non-cardiac chest pain (General disorders) | 9 | 1 | NA | NA
Oedema (General disorders) | 1 | 0 | NA | NA
Oedema peripheral (General disorders) | 2 | 0 | NA | NA
Organ failure (General disorders) | 1 | 0 | NA | NA
Pain (General disorders) | 3 | 0 | NA | NA
Pelvic mass (General disorders) | 1 | 0 | NA | NA
Peripheral swelling (General disorders) | 1 | 0 | NA | NA
Pre-existing condition improved (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 25 | 1 | NA | NA
Stenosis (General disorders) | 1 | 0 | NA | NA
Strangulated hernia (General disorders) | 1 | 0 | NA | NA
Sudden death (General disorders) | 1 | 0 | NA | NA
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | NA | NA
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | NA | NA
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | NA | NA
Biliary colic (Hepatobiliary disorders) | 1 | 0 | NA | NA
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0 | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 5 | 0 | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatic failure (Hepatobiliary disorders) | 4 | 0 | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0 | NA | NA
Hepatitis (Hepatobiliary disorders) | 2 | 0 | NA | NA
Hepatitis acute (Hepatobiliary disorders) | 2 | 0 | NA | NA
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 4 | 0 | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | NA | NA
Jaundice (Hepatobiliary disorders) | 2 | 0 | NA | NA
Liver disorder (Hepatobiliary disorders) | 1 | 0 | NA | NA
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hypersensitivity (Immune system disorders) | 1 | 0 | NA | NA
Abscess intestinal (Infections and infestations) | 1 | 0 | NA | NA
Acute sinusitis (Infections and infestations) | 0 | 1 | NA | NA
Appendicitis perforated (Infections and infestations) | 0 | 1 | NA | NA
Arthritis bacterial (Infections and infestations) | 1 | 0 | NA | NA
Atypical pneumonia (Infections and infestations) | 1 | 0 | NA | NA
Bacterial infection (Infections and infestations) | 1 | 0 | NA | NA
Bartholinitis (Infections and infestations) | 1 | 0 | NA | NA
Biliary sepsis (Infections and infestations) | 1 | 0 | NA | NA
Breast abscess (Infections and infestations) | 1 | 0 | NA | NA
Breast cellulitis (Infections and infestations) | 2 | 0 | NA | NA
Bronchitis (Infections and infestations) | 2 | 0 | NA | NA
COVID-19 (Infections and infestations) | 0 | 5 | NA | NA
COVID-19 pneumonia (Infections and infestations) | 0 | 3 | NA | NA
Cellulitis (Infections and infestations) | 10 | 1 | NA | NA
Cervicitis (Infections and infestations) | 1 | 0 | NA | NA
Chronic tonsillitis (Infections and infestations) | 0 | 1 | NA | NA
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | NA | NA
Colonic abscess (Infections and infestations) | 1 | 0 | NA | NA
Dengue fever (Infections and infestations) | 1 | 0 | NA | NA
Device related infection (Infections and infestations) | 2 | 0 | NA | NA
Ear infection (Infections and infestations) | 1 | 0 | NA | NA
Empyema (Infections and infestations) | 1 | 0 | NA | NA
Encephalitis (Infections and infestations) | 1 | 0 | NA | NA
Erysipelas (Infections and infestations) | 9 | 0 | NA | NA
Escherichia infection (Infections and infestations) | 1 | 0 | NA | NA
Fracture infection (Infections and infestations) | 1 | 0 | NA | NA
Gallbladder empyema (Infections and infestations) | 1 | 0 | NA | NA
Gastroenteritis (Infections and infestations) | 5 | 0 | NA | NA
Gastroenteritis viral (Infections and infestations) | 1 | 0 | NA | NA
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0 | NA | NA
Hepatic infection (Infections and infestations) | 1 | 0 | NA | NA
Hepatitis C (Infections and infestations) | 1 | 0 | NA | NA
Infection (Infections and infestations) | 1 | 0 | NA | NA
Infectious pleural effusion (Infections and infestations) | 1 | 0 | NA | NA
Influenza (Infections and infestations) | 12 | 2 | NA | NA
Intervertebral discitis (Infections and infestations) | 1 | 0 | NA | NA
Kidney infection (Infections and infestations) | 2 | 0 | NA | NA
Liver abscess (Infections and infestations) | 1 | 0 | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | NA | NA
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | NA | NA
Lymphangitis (Infections and infestations) | 3 | 0 | NA | NA
Mastitis (Infections and infestations) | 2 | 0 | NA | NA
Metapneumovirus infection (Infections and infestations) | 1 | 0 | NA | NA
Neutropenic sepsis (Infections and infestations) | 2 | 0 | NA | NA
Otitis media (Infections and infestations) | 1 | 0 | NA | NA
Pneumonia (Infections and infestations) | 35 | 5 | NA | NA
Pneumonia bacterial (Infections and infestations) | 1 | 0 | NA | NA
Pneumonia influenzal (Infections and infestations) | 1 | 0 | NA | NA
Post procedural infection (Infections and infestations) | 2 | 0 | NA | NA
Postoperative wound infection (Infections and infestations) | 2 | 0 | NA | NA
Pulmonary sepsis (Infections and infestations) | 1 | 0 | NA | NA
Pyelonephritis (Infections and infestations) | 3 | 0 | NA | NA
Pyelonephritis acute (Infections and infestations) | 1 | 0 | NA | NA
Respiratory tract infection (Infections and infestations) | 1 | 0 | NA | NA
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | NA | NA
Sepsis (Infections and infestations) | 12 | 0 | NA | NA
Septic shock (Infections and infestations) | 2 | 0 | NA | NA
Sinusitis (Infections and infestations) | 1 | 0 | NA | NA
Skin infection (Infections and infestations) | 1 | 0 | NA | NA
Soft tissue infection (Infections and infestations) | 1 | 0 | NA | NA
Spinal cord infection (Infections and infestations) | 2 | 0 | NA | NA
Staphylococcal infection (Infections and infestations) | 1 | 0 | NA | NA
Streptococcal sepsis (Infections and infestations) | 1 | 0 | NA | NA
Tooth abscess (Infections and infestations) | 1 | 1 | NA | NA
Tooth infection (Infections and infestations) | 1 | 0 | NA | NA
Tracheobronchitis (Infections and infestations) | 1 | 0 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | NA | NA
Urinary tract infection (Infections and infestations) | 17 | 1 | NA | NA
Urosepsis (Infections and infestations) | 5 | 0 | NA | NA
Vascular device infection (Infections and infestations) | 2 | 0 | NA | NA
Viral infection (Infections and infestations) | 2 | 0 | NA | NA
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | NA | NA
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0 | NA | NA
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Fall (Injury, poisoning and procedural complications) | 2 | 1 | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 8 | 2 | NA | NA
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 10 | 0 | NA | NA
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | NA | NA
Inflammation of wound (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Poisoning deliberate (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 4 | 0 | NA | NA
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 0 | NA | NA
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Wound (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 23 | 0 | NA | NA
Aspartate aminotransferase increased (Investigations) | 15 | 0 | NA | NA
Biopsy liver abnormal (Investigations) | 0 | 1 | NA | NA
Blood bilirubin increased (Investigations) | 10 | 0 | NA | NA
Blood creatinine increased (Investigations) | 2 | 0 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | NA | NA
Electrocardiogram abnormal (Investigations) | 1 | 0 | NA | NA
Electrocardiogram change (Investigations) | 1 | 0 | NA | NA
General physical condition abnormal (Investigations) | 3 | 0 | NA | NA
Glomerular filtration rate decreased (Investigations) | 1 | 0 | NA | NA
Haemoglobin decreased (Investigations) | 0 | 1 | NA | NA
Hepatic enzyme increased (Investigations) | 4 | 0 | NA | NA
Mycoplasma test positive (Investigations) | 1 | 0 | NA | NA
Neutrophil count decreased (Investigations) | 6 | 0 | NA | NA
Platelet count decreased (Investigations) | 3 | 0 | NA | NA
SARS-CoV-2 test positive (Investigations) | 0 | 1 | NA | NA
Transaminases increased (Investigations) | 6 | 0 | NA | NA
Waist circumference increased (Investigations) | 1 | 0 | NA | NA
White blood cell count decreased (Investigations) | 1 | 0 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | NA | NA
Food intolerance (Metabolism and nutrition disorders) | 2 | 0 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 8 | 0 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0 | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 0 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Mineral metabolism disorder (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 3 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | NA | NA
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 0 | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 0 | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | NA | NA
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | NA | NA
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | NA | NA
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | NA | NA
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | NA | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | NA | NA
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Altered state of consciousness (Nervous system disorders) | 1 | 0 | NA | NA
Ataxia (Nervous system disorders) | 1 | 0 | NA | NA
Brain oedema (Nervous system disorders) | 1 | 0 | NA | NA
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | NA | NA
Cerebral cyst (Nervous system disorders) | 1 | 0 | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 9 | 1 | NA | NA
Coma (Nervous system disorders) | 1 | 0 | NA | NA
Dizziness (Nervous system disorders) | 4 | 0 | NA | NA
Dysarthria (Nervous system disorders) | 1 | 0 | NA | NA
Dystonia (Nervous system disorders) | 1 | 0 | NA | NA
Encephalopathy (Nervous system disorders) | 1 | 0 | NA | NA
Epilepsy (Nervous system disorders) | 1 | 0 | NA | NA
Facial paresis (Nervous system disorders) | 1 | 0 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | NA | NA
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | NA | NA
Headache (Nervous system disorders) | 7 | 0 | NA | NA
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | NA | NA
Intracranial mass (Nervous system disorders) | 0 | 1 | NA | NA
Ischaemic stroke (Nervous system disorders) | 2 | 0 | NA | NA
Loss of consciousness (Nervous system disorders) | 1 | 0 | NA | NA
Migraine (Nervous system disorders) | 1 | 0 | NA | NA
Neuralgia (Nervous system disorders) | 1 | 0 | NA | NA
Paraesthesia (Nervous system disorders) | 1 | 0 | NA | NA
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 | 0 | NA | NA
Petit mal epilepsy (Nervous system disorders) | 1 | 0 | NA | NA
Sciatica (Nervous system disorders) | 3 | 0 | NA | NA
Seizure (Nervous system disorders) | 3 | 0 | NA | NA
Speech disorder (Nervous system disorders) | 1 | 0 | NA | NA
Spinal cord compression (Nervous system disorders) | 1 | 1 | NA | NA
Syncope (Nervous system disorders) | 6 | 0 | NA | NA
Thalamic infarction (Nervous system disorders) | 1 | 0 | NA | NA
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | NA | NA
Tremor (Nervous system disorders) | 2 | 0 | NA | NA
Device breakage (Product Issues) | 1 | 0 | NA | NA
Device dislocation (Product Issues) | 1 | 0 | NA | NA
Device extrusion (Product Issues) | 1 | 0 | NA | NA
Anxiety (Psychiatric disorders) | 2 | 0 | NA | NA
Apathy (Psychiatric disorders) | 1 | 0 | NA | NA
Confusional state (Psychiatric disorders) | 4 | 0 | NA | NA
Delirium (Psychiatric disorders) | 3 | 0 | NA | NA
Depression (Psychiatric disorders) | 3 | 0 | NA | NA
Mental status changes (Psychiatric disorders) | 1 | 0 | NA | NA
Nervousness (Psychiatric disorders) | 1 | 0 | NA | NA
Suicide attempt (Psychiatric disorders) | 2 | 0 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 12 | 0 | NA | NA
Bladder necrosis (Renal and urinary disorders) | 1 | 0 | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | NA | NA
Haematuria (Renal and urinary disorders) | 1 | 0 | NA | NA
Hydronephrosis (Renal and urinary disorders) | 5 | 0 | NA | NA
Nephritis (Renal and urinary disorders) | 1 | 0 | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 4 | 1 | NA | NA
Prerenal failure (Renal and urinary disorders) | 1 | 0 | NA | NA
Renal colic (Renal and urinary disorders) | 1 | 0 | NA | NA
Renal failure (Renal and urinary disorders) | 2 | 0 | NA | NA
Renal impairment (Renal and urinary disorders) | 1 | 0 | NA | NA
Renal injury (Renal and urinary disorders) | 1 | 0 | NA | NA
Renal tubular disorder (Renal and urinary disorders) | 1 | 0 | NA | NA
Urinary retention (Renal and urinary disorders) | 1 | 0 | NA | NA
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0 | NA | NA
Breast mass (Reproductive system and breast disorders) | 1 | 0 | NA | NA
Breast pain (Reproductive system and breast disorders) | 1 | 0 | NA | NA
Colpocele (Reproductive system and breast disorders) | 1 | 0 | NA | NA
Female genital tract fistula (Reproductive system and breast disorders) | 2 | 0 | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 2 | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 34 | 0 | NA | NA
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | NA | NA
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 19 | 0 | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | NA | NA
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | NA | NA
Menopause (Social circumstances) | 3 | 0 | NA | NA
Postmenopause (Social circumstances) | 0 | 1 | NA | NA
Accelerated hypertension (Vascular disorders) | 1 | 0 | NA | NA
Aortic stenosis (Vascular disorders) | 1 | 0 | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 1 | NA | NA
Embolism (Vascular disorders) | 2 | 0 | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | NA | NA
Jugular vein embolism (Vascular disorders) | 1 | 0 | NA | NA
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | NA | NA
Peripheral ischaemia (Vascular disorders) | 0 | 1 | NA | NA
Phlebitis (Vascular disorders) | 2 | 0 | NA | NA
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | NA | NA
Thrombophlebitis (Vascular disorders) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients- On-treatment Core Phase (N=3246) | All Patients- On-treatment Extension Phase (N=413) | All-patients- Post-treatment Survival Follow-up Core Phase (N=0) | All-patients- Post-treatment Survival Follow-up Extension Phase (N=0)
Anaemia (Blood and lymphatic system disorders) | 597 | 22 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 596 | 23 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 165 | 4 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1981 | 116 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 254 | 13 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 213 | 7 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 216 | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 553 | 11 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 684 | 18 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 237 | 5 | NA | NA
Nausea (Gastrointestinal disorders) | 1160 | 21 | NA | NA
Stomatitis (Gastrointestinal disorders) | 291 | 4 | NA | NA
Vomiting (Gastrointestinal disorders) | 633 | 18 | NA | NA
Asthenia (General disorders) | 627 | 12 | NA | NA
Fatigue (General disorders) | 756 | 14 | NA | NA
Oedema peripheral (General disorders) | 279 | 2 | NA | NA
Pyrexia (General disorders) | 393 | 25 | NA | NA
Nasopharyngitis (Infections and infestations) | 194 | 7 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 191 | 12 | NA | NA
Urinary tract infection (Infections and infestations) | 195 | 16 | NA | NA
Alanine aminotransferase increased (Investigations) | 523 | 10 | NA | NA
Aspartate aminotransferase increased (Investigations) | 456 | 12 | NA | NA
Blood creatinine increased (Investigations) | 199 | 6 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 217 | 3 | NA | NA
Neutrophil count decreased (Investigations) | 623 | 29 | NA | NA
White blood cell count decreased (Investigations) | 336 | 21 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 401 | 7 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 674 | 38 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 426 | 22 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 225 | 9 | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 205 | 1 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 192 | 5 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 263 | 14 | NA | NA
Dizziness (Nervous system disorders) | 235 | 13 | NA | NA
Headache (Nervous system disorders) | 458 | 20 | NA | NA
Insomnia (Psychiatric disorders) | 274 | 2 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 492 | 10 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 275 | 10 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 638 | 4 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 228 | 5 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 431 | 2 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 374 | 6 | NA | NA
Hot flush (Vascular disorders) | 490 | 8 | NA | NA
Hypertension (Vascular disorders) | 227 | 11 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT02941926/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02941926/SAP_001.pdf